CLINICAL TRIAL: NCT05610007
Title: Comparison of Hyperbaric Prilocaine 2% 50 Mg and Hyperbaric Bupivacaine 0.5% 12.5 Mg Against Spinal Anesthesia Recovery Time in Cystoscopy Procedure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes125
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Anesthesia; Reaction
MeSH Terms: interventions — Prilocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prilocaine (Experimental): 50 mg hyperbaric 2% prilocaine (2.5 ml volume) + 25 mcg fentanyl (0.5 ml volume)
  Interventions: Drug: Prilocaine
- bupivacaine (Active Comparator): 12.5, 5 mg hyperbaric 0.5% bupivacaine (2.5 ml volume) + 25 mcg fentanyl (0.5 ml volume)
  Interventions: Drug: Prilocaine

INTERVENTIONS:
Drug: Prilocaine — Patients in the prilocaine group were given 50 mg hyperbaric 2% prilocaine (2.5 ml volume) + 25 mcg fentanyl (0.5 ml volume) before undergoing the cystoscopy procedure.

SUMMARY:
Data regarding the comparison of recovery time from spinal anesthesia between prilocaine and bupivacaine are still relatively limited. The aim of this study was to compare the speed of recovery of spinal anesthesia with hyperbaric prilocaine 2% 50 mg compared to hyperbaric bupivacaine 0.5% 12.5 mg in cystoscopy procedures. By knowing the speed of recovery time, it is hoped that the patient will recover faster, be transferred to the treatment room faster, be safer, and the length of treatment will be shorter so that the quality of service for cystoscopy procedures and patient satisfaction is getting better.

DETAILED DESCRIPTION:
This study is a double-blind randomized clinical trial. This study compared the speed of recovery from spinal anesthesia, as many as 66 subjects were divided into two groups, namely hyperbaric prilocaine 2% 50 mg and hyperbaric bupivacaine 0.5% 12.5 mg who would undergo a cystoscopy procedure. This research was conducted in the urological surgery room of RSCM in January - October 2022, after passing the ethical review and obtaining a location permit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18,
* ASA physical status I - III,
* Normal body mass index according to Quetelet's index,
* Willing to be a research participant and comply with the research rules.

Exclusion Criteria:

* Have a history of allergy to prilocaine or bupivacaine,
* Have a previous history of walking disorders
* Spinal anesthesia is contraindicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 24 hour
  Pain measurement scale felt by patients with a score of 0 = no pain and a score of 10 = unbearable severe pain.

SECONDARY OUTCOMES:
Complication | 24 hour
  Complications that occur due to spinal drug administration, such as chills, hypotension, postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No